CLINICAL TRIAL: NCT04729803
Title: Investigating Attentional Processes: Teleconferencing and Social Anxiety
Brief Title: Attention, Teleconferencing and Social Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000106
Record Dates: First submitted 2020-12-07; First posted 2021-01-29 (Actual); Results first posted 2024-01-08 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Social Anxiety Disorder
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Attention Guidance + Exposure (Experimental): Participants will complete teleconferencing-based exposure trials with an attention guidance component.
  Interventions: Behavioral: Experimental: Attention Guidance + Exposure
- Exposure Alone (Active Comparator): Participants will complete teleconferencing-based exposure trials.
  Interventions: Behavioral: Active Comparator: Exposure Alone
- Attention Control + Exposure (Experimental): Participants will complete teleconferencing-based exposure trials with an attention control component.
  Interventions: Behavioral: Experimental: Attention Control + Exposure

INTERVENTIONS:
Behavioral: Experimental: Attention Guidance + Exposure — 1. Participants will receive a brief standardized psychoeducation module, presented via a video recording.
  2. Participants will then complete up to 10 analogue teleconferencing calls, each lasting a maximum of two minutes.
  3. Between speeches participants will have a 1-minute break.
  4. Participants will complete the subjective units of distress scale (SUDS) before and after each speech trial.
  The experimental attention guidance condition: (1) the intervention rationale will include information about the importance of visually attending to the faces of the audience; (2) participants will be given target audience members to focus their gaze on during the their impromptu response. They will be told that they should look at and focus on the target audience member for the whole response.
  Arms: Attention Guidance + Exposure
Behavioral: Active Comparator: Exposure Alone — 1. Participants will receive a brief standardized psychoeducation module, presented via a video recording.
  2. Participants will then complete up to 10 analogue teleconferencing calls, each lasting a maximum of two minutes.
  3. Between speeches participants will have a 1-minute break.
  4. Participants will complete the subjective units of distress scale (SUDS) before and after each speech trial.
  Arms: Exposure Alone
Behavioral: Experimental: Attention Control + Exposure — 1. Participants will receive a brief standardized psychoeducation module, presented via a video recording.
     F
  2. Participants will then complete up to 10 analogue teleconferencing calls, each lasting a maximum of two minutes. During each call participants will be prompted by one of the audience members.
  3. Between speeches participants will have a 1-minute break.
  4. Participants will complete the subjective units of distress scale (SUDS) before and after each speech trial.
  The experimental attention control condition: (1) the intervention rationale will include information about the importance of attention control; (2) participants will be given target at the center of the screen to focus their gaze on during the their impromptu response. They will be told that they should look at and focus on the target for the whole response.
  Arms: Attention Control + Exposure

SUMMARY:
This study involves completing some online assessments and an intervention for social anxiety that all involve interactions with other people on a teleconferencing call.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75
* Fluent in English because the data collection materials have not yet been standardized in other languages
* Having access to a computer with a webcam and ability to record audio
* Personal Report of Communication Apprehension > 80
* Leibowitz Social Anxiety Scale > 30
* Meets DSM-5 Criteria for Social Anxiety Disorder

Exclusion Criteria:

* Significant visual impairment precluding the use of the eye tracking equipment
* Current, or history of bipolar disorder; current, or history of psychosis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2021-01-18 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratory for the Study of Anxiety Disorders, University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data and analysis syntax will be made available using an open data repository (e.g. osf.io)
Supporting Information: SAP, Analytic Code

RESULTS

PARTICIPANT FLOW:
Groups:
- Attention Guidance + Exposure: Participants will complete teleconferencing-based exposure trials with an attention guidance component.
  Experimental: Attention Guidance + Exposure: 1) Participants will receive a brief standardized psychoeducation module, presented via a video recording.
  2) Participants will then complete up to 10 analogue teleconferencing calls, each lasting a maximum of two minutes.
  3) Between speeches participants will have a 1-minute break. 4) Participants will complete the subjective units of distress scale (SUDS) before and after each speech trial.
  The experimental attention guidance condition: (1) the intervention rationale will include information about the importance of visually attending to the faces of the audience; (2) participants will be given target audience members to focus their gaze on during the their impromptu response. They will be told that they should look at and focus on the target audience member for the whole response.
- Exposure Alone: Participants will complete teleconferencing-based exposure trials.
  Active Comparator: Exposure Alone: 1) Participants will receive a brief standardized psychoeducation module, presented via a video recording.
  2) Participants will then complete up to 10 analogue teleconferencing calls, each lasting a maximum of two minutes.
  3) Between speeches participants will have a 1-minute break. 4) Participants will complete the subjective units of distress scale (SUDS) before and after each speech trial.
- Attention Control + Exposure: Participants will complete teleconferencing-based exposure trials with an attention control component.
  Experimental: Attention Control + Exposure: 1) Participants will receive a brief standardized psychoeducation module, presented via a video recording.
  F 2) Participants will then complete up to 10 analogue teleconferencing calls, each lasting a maximum of two minutes. During each call participants will be prompted by one of the audience members.
  3) Between speeches participants will have a 1-minute break. 4) Participants will complete the subjective units of distress scale (SUDS) before and after each speech trial.
  The experimental attention control condition: (1) the intervention rationale will include information about the importance of attention control; (2) participants will be given target at the center of the screen to focus their gaze on during the their impromptu response. They will be told that they should look at and focus on the target for the whole response.
Period: Overall Study
Arm/Group | Attention Guidance + Exposure | Exposure Alone | Attention Control + Exposure
Started | 13 | 18 | 22
Post-treatment | 7 | 15 | 12
Completed | 6 | 12 | 9
Not Completed | 7 | 6 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Attention Guidance + Exposure | Exposure Alone | Attention Control + Exposure | Total
Number analyzed (Participants) | 13 | 18 | 22 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.20 (1.52) | 18.70 (1.02) | 19.5 (1.77) | 19.13 (1.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 17 | 16 | 46
  Male | 0 | 1 | 6 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 8 | 7 | 20
  Not Hispanic or Latino | 8 | 10 | 15 | 33
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 2 | 6 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 2
  White | 6 | 6 | 8 | 20
  More than one race | 4 | 6 | 3 | 13
  Unknown or Not Reported | 0 | 3 | 4 | 7
Region of Enrollment [Number; unit: participants]
  United States | 13 | 18 | 22 | 53

OUTCOME MEASURES:

1. Primary Outcome: Personal Report of Communication Apprehension Questionnaire
Description: Assessment of communication concerns, range of scores is 24-120; higher scores are worse
Time Frame: prior to the first treatment session, an average of 2 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exposure Alone | Attention Control + Exposure | Attention Guidance + Exposure
Number analyzed (Participants) | 18 | 22 | 13
score on a scale | 88.06 (11.66) | 87.64 (11.91) | 95.69 (14.35)

2. Primary Outcome: Personal Report of Communication Apprehension Questionnaire
Description: Assessment of communication concerns, range of scores is 24-120; higher scores are worse
Time Frame: 1-week follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exposure Alone | Attention Control + Exposure | Attention Guidance + Exposure
Number analyzed (Participants) | 15 | 12 | 7
score on a scale | 70.71 (7.01) | 65.90 (5.36) | 70.00 (1.10)

3. Primary Outcome: Personal Report of Communication Apprehension Questionnaire
Description: Assessment of communication concerns, range of scores is 24-120; higher scores are worse
Time Frame: 2-week follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exposure Alone | Attention Control + Exposure | Attention Guidance + Exposure
Number analyzed (Participants) | 12 | 9 | 6
score on a scale | 70.25 (6.25) | 67.13 (3.23) | 71.00 (1.67)

4. Primary Outcome: Leibowitz Social Anxiety Scale Questionnaire
Description: Assessment of general social anxiety, range of scores is 0-144; higher scores are worse
Time Frame: prior to the first treatment session, an average of 2 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exposure Alone | Attention Control + Exposure | Attention Guidance + Exposure
Number analyzed (Participants) | 18 | 22 | 13
score on a scale | 81.06 (13.40) | 74.50 (13.94) | 87.77 (19.93)

5. Primary Outcome: Leibowitz Social Anxiety Scale Questionnaire
Description: Assessment of general social anxiety, range of scores is 0-144; higher scores are worse
Time Frame: 1-week follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exposure Alone | Attention Control + Exposure | Attention Guidance + Exposure
Number analyzed (Participants) | 15 | 12 | 7
score on a scale | 77.99 (23.60) | 57.70 (19.24) | 71.00 (26.00)

6. Primary Outcome: Leibowitz Social Anxiety Scale Questionnaire
Description: Assessment of general social anxiety, range of scores is 0-144; higher scores are worse
Time Frame: 2-week follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exposure Alone | Attention Control + Exposure | Attention Guidance + Exposure
Number analyzed (Participants) | 12 | 9 | 6
score on a scale | 81.67 (23.52) | 50.13 (15.72) | 71.00 (30.91)

ADVERSE EVENTS:
Time Frame: four weeks
Arm/Group | Exposure Alone | Attention Control + Exposure | Attention Guidance + Exposure
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/22 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/22 | 0/13
Other Adverse Events (participants affected / at risk) | 0/18 | 0/22 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-12-02): https://cdn.clinicaltrials.gov/large-docs/03/NCT04729803/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-05): https://cdn.clinicaltrials.gov/large-docs/03/NCT04729803/SAP_001.pdf
  • Informed Consent Form (2020-12-02): https://cdn.clinicaltrials.gov/large-docs/03/NCT04729803/ICF_002.pdf